CLINICAL TRIAL: NCT00250562
Title: A Multicenter, Double-blind, Randomized, Active Controlled, Parallel Group Trial Comparing the Combinations of Valsartan 80 mg Plus Hydrochlorothiazide 12.5 mg to Valsartan 80 mg in Patients With Mild to Moderate Essential Hypertension Not Adequately Controlled With Valsartan 80mg
Brief Title: A Study in Chinese Mild to Moderate Hypertensive Patients Comparing the Efficacy of Co-Diovan With Diovan.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAH631A2302
Record Dates: First submitted 2005-11-06; First posted 2005-11-08 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2016-11

CONDITIONS: Hypertension
Keywords: Hypertension; Angiotensin II receptor blocker; fixed combination; diuretics
MeSH Terms: conditions — Hypertension | interventions — Valsartan; Hydrochlorothiazide

INTERVENTIONS:
Drug: valsartan plus hydrochlorothiazide

SUMMARY:
Valsartan, an orally active angiotensin II receptor blocker, is registered in most countries worldwide for the treatment of hypertension. In China the usual recommended starting and maintenance dose is 80 mg o.d. The combination of HCTZ 12.5 mg with valsartan 80 mg has been shown to have additive effects in lowering blood pressure compared to valsartan 80 mg in patients not adequately controlled by valsartan 80 mg monotherapy5 or in non-selected patients6. This fixed combination is registered in most countries worldwide.

The potential benefits of these combinations should be evaluated in patients not adequately controlled by valsartan 80 mg monotherapy. This study will compare the efficacy, safety and tolerability of adding HCTZ 12.5 mg to valsartan 80 mg in those hypertensive patients.

This study is not recruiting in the US.

ELIGIBILITY:
Inclusion Criteria:

* - Male or female Outpatients 18 years and older.
* Patients with hypertension defined as the following:
* Newly diagnosed hypertensive patients should have a MSDBP > 95 mmHg and < 110 mmHg.at Visit 1 and 2, Pre-treated hypertensive patients should have a MSDBP > 95 mmHg and < 110 mmHg at Visit 2
* For entrance into the double-blind treatment period (Visit 3), all patients should have a MSDBP of > 90 mmHg and < 110 mmHg
* Patients must have given written informed consent to participate and be willing to participate in the entire study

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1171 (Actual)
Dates: Start 2005-10; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline diastolic blood pressure after 8 weeks

SECONDARY OUTCOMES:
Change from baseline systolic blood pressure after 8 weeks
Diastolic blood pressure less than 90 mmHg or at least a 10 mmHg decrease in diastolic blood pressure after 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceutical, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States

REFERENCES:
- [Result] Sun NL, Zhu JR, Zhao Y, Tu YM; Co-Diovan Trial Investigators. Combination antihypertensive therapy with valsartan and hydrochlorothiazide in Chinese patients with mild-to-moderate hypertension. Curr Med Res Opin. 2008 Oct;24(10):2863-71. doi: 10.1185/03007990802390647. Epub 2008 Aug 29. PMID 18761785